CLINICAL TRIAL: NCT06356896
Title: The Effect of Diaphragmatic Breathing Exercise Applied to Patients Undergoing Coronary Artery Bypass Surgery on Symptom Severity, Sleep Quality and Anxiety.
Brief Title: The Effect of Diaphragmatic Breathing Exercise on Symptom Severity, Sleep Quality and Anxiety in CABG Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Serap Sayar, Asisstant Professor, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023/034
Record Dates: First submitted 2024-03-07; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery; Anxiety; Symptom; Sleep
Keywords: coronary artery bypass; anxiety; symptom; sleep
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Adult patients will be divided into two groups: experimental and control groups. Diaphragmatic breathing exercise will be explained to the patients in the experimental group in the preoperative period. In the preoperative period, the sleep, anxiety and symptom levels of the experimental and control groups will be evaluated.In the post-operative period, the experimental group was reminded to do diaphragmatic breathing exercises on the 2nd, 3rd and 4th days.On the 5th post-operative day, sleep, anxiety and symptom severity of the experimental and control groups will be evaluated.
Who Masked: Participant
Masking Description: Single (Participant) Single Blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental: experimental group (Experimental): Diaphragmatic breathing exercise will be explained practically to the patients in the experimental group in the preoperative period. Anxiety, sleep and symptom levels will be evaluated. 2-3-4 in the post-operative period. On the 5th day, the patient will be encouraged to do diaphragmatic breathing exercises. On the 5th day, anxiety, sleep and symptom levels will be evaluated.
  Interventions: Behavioral: diaphragmatic breathing exercise
- control group (No Intervention): The standard procedure will be applied to the control group without any intervention.

INTERVENTIONS:
Behavioral: diaphragmatic breathing exercise — Each patient's relative should not be in the room, the curtains/screens around the patient bed should be closed, and interventions should be applied in a comfortable environment care will be taken to ensure that the room is quiet and calm. During the first 5 minutes, researchers will explain with pictures how the exercise is done and show it to the patient. The patient will then be asked to perform the exercise for 10 minutes under the supervision of the researchers. If the patient has performed the DBE correctly, the procedure will be discontinued. Otherwise, the patient will be asked to practice for another 5 minutes. If at the end of this period the patient still cannot perform the exercise correctly, he will be removed from the sample. DBE will be performed according to Cleveland Clinic guidelines.
  Arms: experimental: experimental group

SUMMARY:
Coronary artery bypass surgery (CABC) is a commonly performed surgical procedure for the treatment of blockages in the heart vessels. This surgical intervention aims to improve the blood circulation of the patients' heart muscle. However, after CABC, patients may experience symptoms arising from the effect of the operation. These symptoms include shortness of breath, chest pain, sleep problems and a general feeling of restlessness. These symptoms occur as a result of the operation and can limit patients' daily activities, negatively affect their quality of life, and make the rehabilitation process difficult. Diaphragmatic breathing exercise can be an effective strategy for managing symptoms after CABC. This exercise involves deep and controlled breathing and aims to strengthen respiratory muscles, increase lung capacity and improve respiratory efficiency. Diaphragmatic breathing exercise helps breathing occur more efficiently by reducing the movement of the chest wall and can reduce patients' breathing difficulties. Diaphragmatic breathing exercise provides relaxation in the body by calming the sympathetic nervous system and can reduce stress during the sleep process. In this way, patients can experience a deeper and more restful sleep and feel more energetic when they wake up. At the same time, diaphragmatic breathing exercise improves mental state and reduces the effects of stress by providing focus and mental relaxation. This thesis study aims to investigate the effect of diaphragmatic breathing exercise applied to patients undergoing CABC on symptom severity, sleep quality and anxiety. The importance of this study is that it has great potential for managing symptoms after CABC and improving patients' quality of life. Diaphragmatic breathing exercise is expected to be effective in reducing symptoms after CABC, allowing patients to improve their respiratory functions and general health status. Additionally, investigating the effects of this exercise on patients' sleep quality and anxiety may help nurses adopt a more holistic approach in healthcare delivery.

DETAILED DESCRIPTION:
Coronary artery bypass surgery (CABC) is a commonly performed surgical procedure for the treatment of blockages in the heart vessels. This surgical intervention aims to improve the blood circulation of the heart muscle of patients. However, after CABC, patients may experience symptoms arising from the effect of the operation. These symptoms include shortness of breath, chest pain, sleep problems and a general feeling of restlessness. These symptoms occur as a result of the operation and can limit the daily activities of patients, negatively affect their quality of life and make the rehabilitation process difficult.Diaphragmatic breathing exercise can be an effective strategy for managing symptoms after CABC. This exercise involves deep and controlled breathing and aims to strengthen respiratory muscles, increase lung capacity and improve respiratory efficiency.Diaphragmatic breathing exercise helps breathing occur more efficiently by reducing the movement of the chest wall and can reduce patients' breathing difficulties.After CABC, patients' sleep quality can often be negatively affected. Factors such as shortness of breath, pain, discomfort, and time spent in a hospital environment can cause decreases in sleep duration and quality. Sleep disorders can affect patients' rest and recovery processes, reduce their overall quality of life, and prolong the recovery process. Diaphragmatic breathing exercise may be a potential strategy to improve sleep quality. This exercise, which involves deep and controlled breathing as well as relaxation and stress reduction techniques, can improve sleep patterns by promoting relaxation.Diaphragmatic breathing exercise provides relaxation in the body by calming the sympathetic nervous system and can reduce stress during the sleep process. In this way, patients can experience a deeper and more restful sleep and feel more energetic when they wake up.Coronary artery bypass surgery (CABG) is a commonly used surgical method in the treatment of narrowing of the coronary arteries. This surgical procedure aims to improve blood circulation of the heart muscle and improves patients' quality of life. However, increased anxiety levels may be observed in patients undergoing CABG in the postoperative period. This anxiety can affect patients' rehabilitation process and negatively impact their quality of life.Therefore, effective interventions to reduce anxiety in CABG patients are being investigated. Anxiety is a common condition in patients undergoing CABG surgery and may increase in the post-surgical period. This anxiety can be caused by a variety of factors, including physical discomfort, the hospital environment, fear, uncertainty, and concerns about the future. Therefore, it is important to develop an effective intervention to reduce anxiety in CABG patients.Diaphragmatic breathing exercise is a technique used to control breathing and encourage deep breathing. This exercise is known to have positive effects such as reducing stress, providing relaxation and reducing anxiety. Therefore, it is thought that diaphragmatic breathing exercise may have a positive effect on anxiety in CABG patients. This exercise provides relief and relaxation by encouraging the correct use of respiratory muscles. Diaphragmatic breathing exercise involves rhythmically controlling breathing and expanding and contracting the abdominal area. This process helps reduce stress responses by activating the sympathetic nervous system and provide relief by activating the parasympathetic nervous system.The effect of diaphragmatic breathing exercise on anxiety is based on several mechanisms. Breathing deeply and slowly increases the amount of oxygen and reduces the amount of carbon dioxide in the body. This provides relief by reducing the release of cortisol and adrenaline, the body's stress hormones.At the same time, diaphragmatic breathing exercise improves mental state and reduces the effects of stress by providing focus and mental relaxation.This thesis study aims to investigate the effect of diaphragmatic breathing exercise applied to patients undergoing CABC on symptom severity, sleep quality and anxiety. Managing symptoms and improving patients' quality of life after CABC has become an important goal. Research in this field shows that diaphragmatic breathing exercise can reduce symptoms after CABC and reduce patients' general anxiety. However, the information in the literature shows that there are not enough and comprehensive studies on this subject. Therefore, this thesis study aims to evaluate the effect of diaphragmatic breathing exercise on symptom severity, sleep quality and anxiety in patients undergoing CABC. The study is conducted to evaluate the effect of diaphragmatic breathing exercise applied to patients undergoing CABC on symptom severity, sleep quality and anxiety. This study aims to investigate the effectiveness of the care provided by nurses to patients after CABC and its contribution to increasing patient outcomes.The importance of this study is that it has great potential for managing symptoms after CABC and improving patients' quality of life. Diaphragmatic breathing exercise is expected to be effective in reducing symptoms after CABC, allowing patients to improve their respiratory functions and general health status. Additionally, investigating the effects of this exercise on patients' sleep quality and anxiety may help nurses adopt a more holistic approach in healthcare delivery.The findings of this study may offer an effective intervention strategy that can be used in nursing practice in the care of patients after CABC. Diaphragmatic breathing exercise is expected to reduce post-CABC symptoms, improve patients' quality of life, and improve their general anxiety. Nurses can play an important role in implementing this intervention, guiding and supporting patients. Additionally, this study is concerned with identifying an intervention that has the potential to alleviate post-CABC symptoms. Reduction of symptoms, While patients' quality of life increases, their anxiety may decrease. This study has the potential to provide an effective intervention strategy that nurses can use to guide and support patients after CABC.

ELIGIBILITY:
Inclusion Criteria:

* • Being over 18 years old

  * No vision or hearing problems
  * Able to speak and understand Turkish
  * No mental, psychiatric or neurological disabilities
  * Transferred to the clinic on the second postoperative day
  * Those who do not have chronic lung disease (COPD, Asthma, Pulmonary CA.. etc.)
  * Full orientation to person, place and time

Exclusion Criteria:

* If the patient develops any complications during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
cardiovascular surgery symptom inventory | 10 minutes(5th day after surgery)
  It will be applied to adult patients in the intervention and control groups on the 5th post-operative day. Scores between 0 and 140 can be obtained from the inventory. As the scores increase, symptom severity increases.

SECONDARY OUTCOMES:
richards champbell sleep quality scale | 10 minutes(one day before surgery and the 5th day after surgery)
  Patients in the experimental and control groups will be evaluated on the 5th day of pre-op and post-op.A score between "0-25" from the scale indicates very poor sleep, and a score between "76-100" indicates very good sleep. As the scale score increases, the sleep quality of the patients also increases.

OTHER OUTCOMES:
state anxiety inventory | 10 minutes(one day before surgery and the 5th day after surgery)
  It will be applied to the experimental and control groups in the preoperative period and on the 5th post-operative day.A high score on the scale indicates a high level of anxiety; A low score indicates a low level of anxiety.
Personal information form | 2 minutes(one day before surgery)
  Personal information form, literature review as a result, it was created by the researchers. This form contains a total of 11 questions including sociodemographic and descriptive characteristics such as the patient's name and surname, age, gender, marital status, education level, presence of chronic disease, alcohol and cigarette consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Serap SAYAR, PhD, Study Director — KTO Karatay University; Havva Nur YALICI, MSc Student, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The researcher at Konya City Hospital will collect the data.